CLINICAL TRIAL: NCT06736743
Title: Review of Infant Oral Feeding and Skills Study
Brief Title: Review of Infant Oral Feeding and Skills
Acronym: RIOS
Status: Enrolling by invitation | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00120659; AR00057 (Other: Advocate Health)
Record Dates: First submitted 2024-12-10; First posted 2024-12-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Nutrition Disorders; Gastrointestinal Disease; Deglutition Disorder; Feeding Difficulties; Swallowing Difficulties; Humans; Cohort Studies; Infant, Newborn; Infant, Premature, Nutrition; Pediatric Feeding Disorder, Chronic; Retrospective Studies; Breastfeeding; Mental Health Wellness; Intensive Care Units, Neonatal; Bottle Feeding
Keywords: nutrition; infant; neonate; dysphagia; synactive theory of development; life course health development; feeding skill assessment (FSA); SMART Tool; deglutition
MeSH Terms: conditions — Nutrition Disorders; Gastrointestinal Diseases; Deglutition Disorders; Premature Birth; Bronchiolitis Obliterans Syndrome; Breast Feeding; Bottle Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NICU Infants: One cohort of infants who were admitted and discharged during the study period.
  Interventions: Diagnostic Test: SMART Tool for Feeding Skill Assessment

INTERVENTIONS:
Diagnostic Test: SMART Tool for Feeding Skill Assessment — Infant Oral Feeding Skill Assessment (FSA) done using SMART Tool

SUMMARY:
This study evaluates the infant's feeding skill level at discharge from the neonatal intensive care unit. The goal is to determine whether the ability to "full feed by volume" implies "full skill development" for infant oral feeding.

DETAILED DESCRIPTION:
Situation: Feeding Problems in Infancy

Feeding problems are a frequent complication for infants in the neonatal intensive care unit (NICU), with an estimated 80% of infants experiencing feeding difficulties during their NICU stay. Inadequate oral feeding (by volume) is one of the most common reasons for prolonged NICU stays. Feeding problems are common reasons for hospital readmission in the moderate and late preterm population. In a large multicenter retrospective study of premature infants born before 33 weeks gestation, less than 4% were discharged from NICU with feeding tubes (nasogastric or gastrostomy) for severe feeding problems. However, in the pediatric setting, a meta-analysis found that 42% of premature infants born before 37 weeks had ongoing feeding problems before four years of age. The 10x difference in the prevalence of feeding problems in NICU and pediatric settings implies that infants either have inadequate feeding skills at discharge or develop them later at home. The disparity in the literature begs the question of whether clinicians are adequately assessing feeding skill development in the NICU setting.

In severe cases, feeding problems in childhood cause immense stress to the child and family at mealtime. Pediatric Feeding Disorder (PFD) is defined as impaired oral intake that is not age-appropriate and is associated with medical, nutritional, feeding skills, and/or psychosocial dysfunction. While a skill-based approach to treating PFD is essential in the pediatric world, skill-based information is not fully appreciated in the NICU.

Background: Skill Based Feeding

Feeding management is central to the baby's physiological balance, growth, behavioral display of pleasure, and a nurturing relationship with the parent. The acquisition of safe and efficient nipple-feeding skills is a complex task and one of the most challenging milestones for most preterm or high-risk infants to achieve. Premature infants are at higher risk of feeding problems compared to term infants due to 1. Innate differences in muscle tone, state regulation, endurance, and suck-swallow-breathing coordination; 2. Disruption of in utero brain development due to decreased myelination and white matter disturbances, and 3. They have higher nutritional requirements per kilogram body weight than term infants and are less tolerant of high fluid volumes. Similarly, full-term infants with complex conditions and syndromes may have altered anatomy, physiology and neurodevelopment, which impact oral feeding.

Cue-based feeding (CBF) is considered best practice as infants transition to independent oral feeding skills. Cue-based feeding is a method that combines the use of non-nutritive sucking (NNS) to promote awake behavior for feeding, the use of behavioral assessment to identify readiness for feeding, and systematic observation of and response to infant behavior cues to regulate frequency, duration, and volume of oral feedings. CBF has been shown to have several benefits, such as earlier transition to oral feedings, reduced length of stay, improved physiological maturity, improved nutritional intake, and reduced stress on the family.

A wide range of infant feeding skill assessment tools exist; however, no gold-standard tool has been identified in the literature due to inadequate psychometric tests and feasibility. The study team developed an infant oral feeding skill assessment tool called the SMART Tool, which provides a numerical score before and after feed. The SMART tool evaluates feeding skills across five domains: State of arousal, motor tone, autonomic instability, response to stimulation, and total oral skills. These domains form the acronym of SMART Tool. The Synactive Theory of Development provided the theoretical basis for the SMART tool's design and also aligns with trauma-informed care principles, neonatal integrative developmental care model, life course health development intervention, and infant-family-centered developmental care. The post-feed SMART Tool score classifies the infant feeding skills into three categories: caution (25 to 60), developing (60 to 90), and capable (91 to 100). The SMART tool was designed to meet the needs of NICU clinicians, providing an objective measure of the safety and quality of feedings that can replace the traditional volume-driven approach. The SMART Tool was prospectively tested in four Level III Neonatal Intensive care units (NICU) in the Advocate Health system and shown to be valid and reliable for infant feeding skill assessment. This tool has been integrated into daily clinical usage at 15 NICUs within Advocate Health.

Analysis:

No neonatal feeding skill assessment at Discharge Historically, there has been a focus on the quantity (volume) of oral intake versus the quality (skill). The American Academy of Pediatrics requires "oral feeding sufficient to support appropriate growth" for infants as part of its criterion for hospital discharge. (American Academy of Pediatrics Committee on & Newborn, 2008) This criterion perpetuates the focus on volume rather than skill for infant feeding in the NICU.

Clinicians' most significant assumption is that if an infant can complete oral feedings by volume, the infant is developmentally mature and has adequate feeding skills. No universal policy measures the infant's oral feeding skill level at discharge. The study team believes this is essential information for parents and pediatricians to know about infants' feeding skills, like hearing tests or heart screening. The study team believes that every neonatal discharge summary from the NICU should communicate the infant's feeding skill level to outpatient pediatricians so that they can monitor it closely. Doing so provides continuity of care about the safety and quality of feeds.

Plan: Evaluate skills at discharge

In this pilot retrospective study, the study team intends to evaluate the legitimacy of the assumption that if an infant can complete oral feedings by volume, the infant demonstrates mature, capable feeding skills. SMART Tool qualifies the oral feeding skill level as "caution," "developing," and "capable." If the assumption is valid, all infants with full oral feeds at discharge should be in the "capable" category. The first aim is to check if any infants were in the "caution" or "developing" categories at discharge. The second aim is to describe the distribution of feeding skills levels at discharge.

This study's most powerful impact is dispelling the assumption that "full oral feeds" are the same as "full skill development." This will be pilot data to enable us to do a prospective multicenter study to recheck this assumption on a larger dataset and categorize the feeding level in different situations.

In the future, this study can help us with two big impacts - 1. Change national policy on infant discharge to include some concepts of feeding quality, and 2. Identify those at risk of future pediatric feeding disorders earlier and monitor meaningful outcomes for family and society.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted and discharged from Advocate Illinois Masonic Medical Center (AIMMC) Neonatal Intensive Care Unit (NICU) from April 1, 2024 to September 30, 2024

Exclusion Criteria:

* Discharged without attaining full independent oral feeds by volume. This excludes infant deaths and transfers without attaining full oral feeds.

Ages: 22 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates admitted and discharged from Advocate Illinois Masonic Medical Center (AIMMC) Neonatal Intensive Care Unit (NICU)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Capable Feeding Skills at Discharge | At discontinuation of SMART Tool Scoring for up to 6 months.
  Based on the Last Feeding Skill Assessment (FSA) Score, calculate the percentage of infants in the "capable" range/ total included infants.
  The SMART tool evaluates feeding skills across five domains: State of arousal, motor tone, autonomic instability, response to stimulation, and total oral skills. The score has a minimum value of 25 and a maximum value of 100; higher scores mean a better outcome. The post-feed SMART Tool score classifies the infant feeding skills into three categories: caution (25 to 60), developing (60 to 90), and capable (91 to 100).

SECONDARY OUTCOMES:
Feeding Skills Distribution at Discharge. | At discontinuation of SMART Tool Scoring for up to 6 months.
  Based on the Last Feeding Skill Assessment (FSA) Score, show the distribution of infant feeding levels in three categories: caution, developing, and capable. The SMART tool evaluates feeding skills across five domains: State of arousal, motor tone, autonomic instability, response to stimulation, and total oral skills. The score has a minimum value of 25 and a maximum value of 100; higher scores mean a better outcome. The post-feed SMART Tool score classifies the infant feeding skills into three categories: caution (25 to 60), developing (60 to 90), and capable (91 to 100).

OTHER OUTCOMES:
Last FSA Score at discontinuation of SMART Tool scoring. | At discontinuation of SMART Tool Scoring for up to 6 months.
  Last Feeding Skill Assessment (FSA) Score when SMART Tool scoring was discontinued as per NICU policy.
  The SMART tool evaluates feeding skills across five domains: State of arousal, motor tone, autonomic instability, response to stimulation, and total oral skills. The score has a minimum value of 25 and a maximum value of 100; higher scores mean a better outcome. The post-feed SMART Tool score classifies the infant feeding skills into three categories: caution (25 to 60), developing (60 to 90), and capable (91 to 100).
Length of Stay | Duration of hospitalization in days, for up to 6 months.
  Length of Stay in Hospital
Time from Start oral feeds to Full oral feeds | From start of oral feeds to removal of Nasogastric tubes in days, for up to 6 months.
  Days from initiation of oral feeds to discontinuing nasogastric tube.
Breastfeeding at Discharge | At discharge from the hospital for up to 6 months.
  Percentage of infants with any direct breastfeeding at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Mishra, MD, FAAP, Principal Investigator — Advocate Health
Locations (1):
- Advocate Illinois Masonic Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanders MR, Hall SL. Trauma-informed care in the newborn intensive care unit: promoting safety, security and connectedness. J Perinatol. 2018 Jan;38(1):3-10. doi: 10.1038/jp.2017.124. Epub 2017 Aug 17. PMID 28817114
- [Background] Russ SA, Hotez E, Berghaus M, Verbiest S, Hoover C, Schor EL, Halfon N. What Makes an Intervention a Life Course Intervention? Pediatrics. 2022 May 1;149(Suppl 5):e2021053509D. doi: 10.1542/peds.2021-053509D. PMID 35503318
- [Background] Pineda R, Prince D, Reynolds J, Grabill M, Smith J. Preterm infant feeding performance at term equivalent age differs from that of full-term infants. J Perinatol. 2020 Apr;40(4):646-654. doi: 10.1038/s41372-020-0616-2. Epub 2020 Feb 17. PMID 32066844
- [Background] Goday PS, Huh SY, Silverman A, Lukens CT, Dodrill P, Cohen SS, Delaney AL, Feuling MB, Noel RJ, Gisel E, Kenzer A, Kessler DB, Kraus de Camargo O, Browne J, Phalen JA. Pediatric Feeding Disorder: Consensus Definition and Conceptual Framework. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):124-129. doi: 10.1097/MPG.0000000000002188. PMID 30358739
- [Background] Browne JV, Jaeger CB, Kenner C; Gravens Consensus Committee on Infant and Family Centered Developmental Care. Executive summary: standards, competencies, and recommended best practices for infant- and family-centered developmental care in the intensive care unit. J Perinatol. 2020 Sep;40(Suppl 1):5-10. doi: 10.1038/s41372-020-0767-1. PMID 32859958
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn. Hospital discharge of the high-risk neonate. Pediatrics. 2008 Nov;122(5):1119-26. doi: 10.1542/peds.2008-2174. PMID 18977994
- [Background] Alshaikh B, Yusuf K, Dressler-Mund D, Mehrem AA, Augustine S, Bodani J, Yoon E, Shah P; Canadian Neonatal Network (CNN) and Canadian Preterm Birth Network (CPTBN) Investigators. Rates and Determinants of Home Nasogastric Tube Feeding in Infants Born Very Preterm. J Pediatr. 2022 Jul;246:26-33.e2. doi: 10.1016/j.jpeds.2022.03.012. Epub 2022 Mar 14. PMID 35301017
- [Background] Milette I, Martel MJ, Ribeiro da Silva M, Coughlin McNeil M. Guidelines for the Institutional Implementation of Developmental Neuroprotective Care in the Neonatal Intensive Care Unit. Part A: Background and Rationale. A Joint Position Statement From the CANN, CAPWHN, NANN, and COINN. Can J Nurs Res. 2017 Jun;49(2):46-62. doi: 10.1177/0844562117706882. PMID 28841058
- [Background] Edwards L, Cotten CM, Smith PB, Goldberg R, Saha S, Das A, Laptook AR, Stoll BJ, Bell EF, Carlo WA, D'Angio CT, DeMauro SB, Sanchez PJ, Shankaran S, Van Meurs KP, Vohr BR, Walsh MC, Malcolm WF; Eunice Kennedy Shriver National Institute of Child Health and Human Development. Inadequate oral feeding as a barrier to discharge in moderately preterm infants. J Perinatol. 2019 Sep;39(9):1219-1228. doi: 10.1038/s41372-019-0422-x. Epub 2019 Jul 11. PMID 31296918
- [Background] Lubbe W. Clinicians guide for cue-based transition to oral feeding in preterm infants: An easy-to-use clinical guide. J Eval Clin Pract. 2018 Feb;24(1):80-88. doi: 10.1111/jep.12721. Epub 2017 Mar 2. PMID 28251754
- [Background] Pados BF, Hill RR, Yamasaki JT, Litt JS, Lee CS. Prevalence of problematic feeding in young children born prematurely: a meta-analysis. BMC Pediatr. 2021 Mar 6;21(1):110. doi: 10.1186/s12887-021-02574-7. PMID 33676453